CLINICAL TRIAL: NCT00867308
Title: Phase II Trial of High Dose Lenalidomide in Patients With MDS and AML With Trilineage Dysplasia (AML-TLD)
Brief Title: Trial of High Dose Lenalidomide in Patients With MDS and AML With Trilineage Dysplasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0882; RV- MDS-PI-295 (Other: Celgene Corporation); NA_00019818 (Other: JHMIRB)
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Myelodysplastic Syndrome
Keywords: IPSS Int-2; high risk myelodysplastic syndrome; MDS); 5q31.1 deletions
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lenalidomide 15 mg (Experimental): Patients diagnosed with high risk Myelodysplastic syndrome (MDS), regardless of 5q deletion status, will receive lenalidomide 15 mg per day orally, on days 1-28 of a 42 day cycle for 2 cycles. At this point, patients meeting protocol specified response criteria will proceed to Continuing Therapy on a reduced dose of lenalidomide until progression.
  Patients not achieving response will receive 2 additional cycles of treatment, whereupon response will again be assessed. Patients achieving response at this point will proceed to Continuing Therapy as described.
  Patients without evidence of response after 4 cycles will be taken off-study.
  Interventions: Drug: Lenalidomide 15 mg
- Lenalidomide 50 mg (Experimental): Patients diagnosed with high risk Myelodysplastic syndrome (MDS), regardless of 5q deletion status, will receive lenalidomide 50 mg per day orally, on days 1-28 of a 42 day cycle for 2 cycles. At this point, patients meeting protocol specified response criteria will proceed to Continuing Therapy on a reduced dose of lenalidomide until progression.
  Patients not achieving response will receive 2 additional cycles of treatment, whereupon response will again be assessed. Patients achieving response at this point will proceed to Continuing Therapy as described.
  Patients without evidence of response after 4 cycles will be taken off-study.
  Interventions: Drug: Lenalidomide 50 mg

INTERVENTIONS:
Drug: Lenalidomide 50 mg
  Other Names: Revlimid
  Arms: Lenalidomide 50 mg
Drug: Lenalidomide 15 mg
  Other Names: Revlimid
  Arms: Lenalidomide 15 mg

SUMMARY:
This is a phase II study of lenalidomide in patients with myelodysplastic syndrome (MDS) and with acute myeloid leukemia (AML) with trilineage dysplasia. Patients will receive two cycles of lenalidomide. Patients who respond may given additional cycles of lenalidomide until disease progression.

DETAILED DESCRIPTION:
This is a single center open label phase II study of lenalidomide in IPSS Int-1 with increased blasts or hematologic needs with 5q31.1 deletions who have failed to respond to standard dose lenalidomide., IPSS Int-1 with increased blasts or hematologic needs without 5q31.1 deletions, and Int-2 and high risk myelodysplastic syndrome (MDS) patients with or without 5q31.1 deletions, regardless of whether they have received lenalidomide previously or not. Patients will receive two cycles of 15 mg daily lenalidomide (later amended to 50 mg daily lenalidomide) given on days 1-28 out of a 42 day cycle. Within each of the two cycles of lenalidomide, patients will be given up to three weeks with no drug treatment to recover. Patients who fail to respond after two cycles of treatment may receive two additional cycles if stable. Patients who develop clinical response may continue to receive drug until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* MDS or MDS/AML
* Patients must not have received any other treatment for their disease, including hematopoietic growth factors, within three weeks of beginning the trial
* ECOG performance status of 0, 1, or 2 at study entry
* All study participants must be registered into the mandatory REMS® program, and be willing and able to comply with the requirements of RevAssist®.
* Patients must have no clinical evidence of CNS or pulmonary leukostasis, disseminated intravascular coagulation, or CNS leukemia.
* Subjects must agree to use appropriate contraception.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 21 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide except for MDS patients with del 5q31.1 abnormalities..
* Concurrent use of other anti-cancer agents or treatments.
* Patients may not have received prior AML induction chemotherapy or stem cell transplant. However, patients with secondary MDS who have received a stem cell transplant for other indications (eg lymphoma, multiple myeloma) will be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy DeZern, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zeidan AM, Smith BD, Carraway HE, Gojo I, DeZern A, Gore SD. A phase 2 trial of high dose lenalidomide in patients with relapsed/refractory higher-risk myelodysplastic syndromes and acute myeloid leukaemia with trilineage dysplasia. Br J Haematol. 2017 Jan;176(2):241-247. doi: 10.1111/bjh.14407. Epub 2016 Oct 28. PMID 27790720

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants on the 15mg arm and 3 participants on the 50mg arm were screen failures.
Period: Overall Study
Arm/Group | Lenalidomide 15 mg | Lenalidomide 50 mg
Started | 9 | 18
Completed | 0 | 0
Not Completed | 9 | 18
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 4
Not completed — Lack of Efficacy | 6 | 12
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide 15 mg | Lenalidomide 50 mg | Total
Number analyzed (Participants) | 9 | 18 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 6 | 14 | 20
Age, Continuous [Median (Full Range); unit: years] | 77 [47 to 88] | 70 [53 to 79] | 72 [47 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 8 | 14 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Number of participants with a complete or partial response according to International Working Group 2006 criteria.
Time Frame: 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide 15 mg | Lenalidomide 50 mg
Number analyzed (Participants) | 9 | 18
Participants
  Complete response | 0 | 0
  Partial response | 0 | 2

2. Secondary Outcome: Grade 3-4 Toxicity
Description: Number of participants who experienced at least one grade 3-4 non-hematological toxicity by CTCAE 3.0 that was attributed to lenalidomide.
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide 15 mg | Lenalidomide 50 mg
Number analyzed (Participants) | 9 | 18
Participants | 6 | 12

ADVERSE EVENTS:
Time Frame: Up to 8 months
Description: Due to significant cytopenias in all participants at presentation and throughout the trial, hematologic toxicity was only reported where bone marrow aplasia lasted for >3 weeks from last dose of lenalidomide with a bone marrow cellularity of <5% without evidence of leukemia. Adverse events were collected weekly throughout the trial.
Arm/Group | Lenalidomide 15 mg | Lenalidomide 50 mg
All-Cause Mortality (participants affected / at risk) | 3/9 | 2/18
Serious Adverse Events (participants affected / at risk) | 3/9 | 9/18
Other Adverse Events (participants affected / at risk) | 7/9 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide 15 mg (N=9) | Lenalidomide 50 mg (N=18)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Weakness - leg (Nervous system disorders) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 1 (1) | 1 (1)
Fungal pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Pericarditis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide 15 mg (N=9) | Lenalidomide 50 mg (N=18)
Anemia (Investigations) | 2 (2) | 0 (0)
Anorexia (General disorders) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Bleeding (Blood and lymphatic system disorders) | 3 (3) | 3 (5)
Bruising (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Confusion (Nervous system disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 6 (8)
Cough (General disorders) | 3 (3) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Edema (Cardiac disorders) | 1 (1) | 7 (10)
Epistaxis (Blood and lymphatic system disorders) | 4 (5) | 3 (3)
Fatigue (General disorders) | 5 (5) | 8 (12)
Febrile neutropenia (Infections and infestations) | 3 (3) | 1 (1)
Fever (Infections and infestations) | 1 (2) | 2 (2)
Hallucination (Nervous system disorders) | 0 (0) | 2 (2)
Headache (General disorders) | 1 (2) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Hoarseness (General disorders) | 0 (0) | 2 (2)
Hyperbilirubinemia (Investigations) | 2 (2) | 1 (1)
Hypokalemia (Investigations) | 1 (1) | 1 (1)
Hyponatremia (Investigations) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 2 (2) | 0 (0)
Lightheadedness (Cardiac disorders) | 0 (0) | 2 (2)
Myalgia (General disorders) | 0 (0) | 6 (11)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Pain - back (General disorders) | 0 (0) | 2 (2)
Pain - chest (General disorders) | 1 (1) | 1 (1)
Pain - tooth (General disorders) | 0 (0) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2) | 8 (13)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 6 (9)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Thrombocytopenia (Investigations) | 3 (3) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Weakness (Nervous system disorders) | 0 (0) | 6 (6)
Xerosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Xerostomia (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes